CLINICAL TRIAL: NCT00872599
Title: The Effect of a PPAR Alpha Agonist on CYP Monooxygenase Activity in Humans
Brief Title: The Effect of a Peroxisome Proliferator-activated Receptor (PPAR) Alpha Agonist on Cytochrome P450 (CYP) Monooxygenase Activity in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PPAR Alpha Agonist; Grant# DK38226-21
Record Dates: First submitted 2009-03-26; First posted 2009-03-31 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension
Keywords: Hypertension; Phenotyping; High Salt intake; frequently sampled IV glucose tolerance test(FSIVGTT); fenofibrate; epoxyeicosatrienoic acids; hydroxyeicosatetraenoic acids; dihydroxyeicosatrienoic acid; PPAR Alpha Agonist; CYP Monooxygenase Activity
MeSH Terms: conditions — Hypertension | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo, then fenofibrate (Placebo Comparator): Randomized study of fenofibrate versus placebo during high salt diet
  Interventions: Drug: fenofibrate; Drug: Placebo
- Fenofibrate, then placebo (Placebo Comparator): Randomized study of fenofibrate versus placebo during high salt intake.
  Interventions: Drug: fenofibrate; Drug: Placebo

INTERVENTIONS:
Drug: fenofibrate — Subjects will be randomized to receive either fenofibrate 160 mg/day or matching placebo for five days by mouth.
  Other Names: Tricor
Drug: Placebo — Subjects will be randomized to receive placebo or fenofibrate for five days by mouth

SUMMARY:
The hypothesis is to test to see if the drug fenofibrate will increase important chemicals in the body and specifically in the kidney, help to rid the body of salt by the kidneys, decrease blood pressure and improve insulin sensitivity during high-salt intake in individuals with hypertension.

DETAILED DESCRIPTION:
Hypertension affects 73 million people in the United States and a billion people worldwide and contributes to death due to stroke, myocardial infarction, end-stage kidney disease and congestive heart failure. Fifty to 60% of individuals with hypertension have "salt-sensitive" hypertension, characterized by an exaggerated blood pressure response to increased salt intake. Salt-sensitive hypertension is associated with increased mortality due to cardiovascular disease.

This study will test the hypothesis that administration of a PPARa agonist, an intervention increases renal tubular Cyp2c and 4a expression in rodents, will increase urinary excretion of 20-hydroxyeicosatetraenoic acid(HETE) and epoxyeicosatrienoic acids(EET)s, induce natriuresis, decrease blood pressure, and improve insulin sensitivity during high-salt intake in individuals with hypertension.

Metabolites of the P450 arachidonic acid monooxygenases play an important role in the regulation of blood pressure in rodent models.

Targeted disruption of murine Cyp4a genes provides insight into the roles of renal monooxygenases and epoxygenases in the regulation of salt excretion and blood pressure.

PPARa agonists induce the expression of renal tubular monoxygenases and epoxygenases and decrease blood pressure in both Ang II- dependent and salt-sensitive rodent models of hypertension.

PPARa agonists have been reported to reduce blood pressure in clinical trials in humans. The effect of PPARa agonist on renal vasodilation, sodium excretion and excretion of urinary epoxygenase or monooxygenase products in response to salt loading is not known.

The regulation of urinary 20-HETE excretion may be impaired in human hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory subjects, 18-70 years of age, inclusive
* For female subjects, the following conditions must be met Postmenopausal status for at least 1 year, or Status post surgical sterilization, or If of childbearing potential, utilization of adequate birth control and willingness to undergo urine beta-hcg testing prior to drug treatment and on every study day

Exclusion Criteria:

* Secondary causes of hypertension
* Diabetes type 1 or type 2 as defined by a fasting glucose of 126 mg/dl or greater or the use of anti-diabetic medication
* Use of hormone replacement therapy
* Statin or fibrate therapy
* A seated systolic blood pressure(SBP) greater than 179 mmHg or a seated diastolic blood pressure(DBP) greater than 110 mmHg
* Pregnancy
* Breast-feeding
* Cardiovascular disease such as history of myocardial infarction, presence of angina pectoris, significant arrhythmia, congestive heart failure, (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
* Treatment with anticoagulants
* History of serious neurologic diseases such as cerebral hemorrhage,stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Diagnosis of asthma
* Clinically significant gastrointestinal impairment that could interfere with drug absorption
* Impaired hepatic function (aspartate aminotransferase [AST] and or alanine aminotransferase [ALT] > 2.0 x upper range)
* Known preexisting gallbladder disease
* Impaired renal function (eGFR < 60 ml/min/1.73M2)
* Hematocrit < 35%
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Treatment with a glucocorticoid therapy
* Treatment with lithium salts
* History of of alcohol or drug abuse
* Treatment with any investigational drug in the 1 month preceding the study
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
* Inability to comply with the protocol, e.g uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Gilbert K, Nian H, Yu C, Luther JM, Brown NJ. Fenofibrate lowers blood pressure in salt-sensitive but not salt-resistant hypertension. J Hypertens. 2013 Apr;31(4):820-9. doi: 10.1097/HJH.0b013e32835e8227. PMID 23385647
- [Derived] Ramirez CE, Shuey MM, Milne GL, Gilbert K, Hui N, Yu C, Luther JM, Brown NJ. Arg287Gln variant of EPHX2 and epoxyeicosatrienoic acids are associated with insulin sensitivity in humans. Prostaglandins Other Lipid Mediat. 2014 Oct;113-115:38-44. doi: 10.1016/j.prostaglandins.2014.08.001. Epub 2014 Aug 28. PMID 25173047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After providing informed consent, subjects underwent a history and physical examination, screening electrocardiogram and laboratory assessment. Subjects were excluded if they did not meet inclusion and exclusion criteria.
Pre-assignment Details: All anti-hypertensive medications were discontinued for 3 weeks. Participants who met blood pressure safety criteria were discontinued. Remaining participants underwent a 6-day low salt diet period and study day prior to randomization. Thirty-three of 75 enrolled met inclusion criteria, and were not withdrawn for high blood pressure during washout.
Groups:
- Placebo, Then Fenofibrate: Subjects underwent two consecutive high salt (200mmol/d) periods. During the first they received matching placebo. During the second they received fenofibrate 160mg/d.
- Fenofibrate, Then Placebo: Subjects underwent two consecutive high salt (200mmol/d) periods. During the first they received fenofibrate 160mg/d. During the second they received matching placebo.
Period: First Washout Period After Low Salt
Arm/Group | Placebo, Then Fenofibrate | Fenofibrate, Then Placebo
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: First Drug During High Salt Intake
Arm/Group | Placebo, Then Fenofibrate | Fenofibrate, Then Placebo
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Second Washout Period
Arm/Group | Placebo, Then Fenofibrate | Fenofibrate, Then Placebo
Started | 16 | 17
Completed | 15 | 16
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Second Drug During High Salt Intake
Arm/Group | Placebo, Then Fenofibrate | Fenofibrate, Then Placebo
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number who completed the screening and low salt diet and were randomized.
Arm/Group | Study Group
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure During High Salt Intake and Fenofibrate Treatment Compared to High Salt Intake and Placebo Treatment
Description: Difference in blood pressure (mean arterial pressure) measured on the last day of high salt intake and fenofibrate treatment minus blood pressure (mean arterial pressure) measured during high salt intake and placebo treatment in participants classified as being salt-sensitive versus salt-resistant.
  Participants were classified as salt-sensitive if the average study day mean arterial pressure (MAP) was at least 5 mmHg higher during the high salt placebo arm than during low salt intake.
Time Frame: pressure measured on day 6 of high salt fenofibrate minus pressure measured on day 6 of high salt placebo
Population: All subjects who completed entire protocol
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Salt-resistant Hypertension: Subjects whose average study day mean arterial pressure was less than 5 mmHg higher during high salt intake compared to low salt intake
- Salt-sensitive Hypertension: Subjects were classified as salt-sensitive if the average study day mean arterial pressure was at least 5 mmHg higher during high salt placebo compared to low salt intake
Arm/Group | Salt-resistant Hypertension | Salt-sensitive Hypertension
Number analyzed (Participants) | 17 | 14
mm Hg | 2.0 (7.1) | -3.4 (6.5)

2. Secondary Outcome: HDL-cholesterol Measured During High Salt Fenofibrate in Salt-resistant and Salt-sensitive Hypertension
Description: HDL-cholesterol concentration measured on the last day of fenofibrate treatment in salt-resistant and salt-sensitive hypertensive patients
Time Frame: Measured on day 6 of high salt intake and fenofibrate treatment
Population: All subjects who completed the protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Salt-resistant Hypertension | Salt-sensitive Hypertension
Number analyzed (Participants) | 17 | 14
mg/dL | 54.1 (20) | 52.1 (15.8)

ADVERSE EVENTS:
Arm/Group | Placebo | Fenofibrate
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 2/33 | 2/33
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | Fenofibrate (N=33)
IV infiltration or bruising (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
High blood pressure during washout phase (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No